CLINICAL TRIAL: NCT00700817
Title: The Effect of Liraglutide Compared to Sitagliptin, Both in Combination With Metformin in Subjects With Type 2 Diabetes. A 26-week, Randomised, Open-label, Active Comparator, Three-armed, Parallel-group, Multi-centre, Multinational Trial With a 52-week Extension
Brief Title: The Effect of Liraglutide Compared to Sitagliptin, Both in Combination With Metformin on Glycaemic Control in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1860; 2007-003937-17 (EudraCT Number)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg (Experimental): Once-daily subcutaneous dose of liraglutide 1.2 mg with at least 1500 mg metformin/day (tablets) for 26 weeks. First week for up-titration of liraglutide from 0.6 mg to 1.2 mg. Subjects continued to receive liraglutide 1.2 mg once daily in extension period 1 (weeks 26-52) and extension period 2 (weeks 52-78).
  Interventions: Drug: liraglutide; Drug: metformin
- Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg (Experimental): Once-daily subcutaneous dose of liraglutide 1.8 mg with at least 1500 mg metformin/day (tablets) for 26 weeks. First 2 weeks for up-titration of liraglutide from 0.6 mg to 1.8 mg. Subjects continued to receive liraglutide 1.8 mg once daily in extension period 1 (weeks 26-52) and extension period 2 (weeks 52-78).
  Interventions: Drug: metformin; Drug: liraglutide
- Sita -> Sita (Active Comparator): Once-daily dose of sitagliptin 100 mg (tablets) with at least 1500 mg metformin/day (tablets) for 26 weeks. Subjects continued to receive 100 mg sitagliptin once daily in extension period 1 (weeks 26-52).
  Interventions: Drug: sitagliptin; Drug: metformin
- Sita -> Sita -> Lira 1.2 mg (Experimental): Once-daily dose of sitagliptin 100 mg (tablets) with at least 1500 mg metformin/day (tablets) for 26 weeks. Subjects continued to receive 100 mg sitagliptin once daily in extension period 1 (weeks 26-52). In extension period 2 (weeks 52-78), subjects were randomised to liraglutide 1.2 mg + metformin.
  Interventions: Drug: liraglutide; Drug: sitagliptin; Drug: metformin
- Sita -> Sita -> Lira 1.8 mg (Experimental): Once-daily dose of sitagliptin 100 mg (tablets) with at least 1500 mg metformin/day (tablets) for 26 weeks. Subjects continued to receive 100 mg sitagliptin once daily in extension period 1 (weeks 26-52). In extension period 2 (weeks 52-78), subjects were randomised to liraglutide 1.8 mg + metformin.
  Interventions: Drug: sitagliptin; Drug: metformin; Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — 1.2 mg once daily, subcutaneous (under the skin) injection
  Arms: Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg; Sita -> Sita -> Lira 1.2 mg
Drug: sitagliptin — Tablets, 100 mg daily
  Arms: Sita -> Sita; Sita -> Sita -> Lira 1.2 mg; Sita -> Sita -> Lira 1.8 mg
Drug: metformin — Tablets, minimum 1500 mg daily
Drug: liraglutide — 1.8 mg once daily, subcutaneous (under the skin) injection
  Arms: Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg; Sita -> Sita -> Lira 1.8 mg

SUMMARY:
This trial is conducted in Europe and North America. The aim of this trial is to compare the effect on blood sugar control of liraglutide or sitagliptin, both in combination with metformin, in subjects with type 2 diabetes inadequately controlled with metformin alone.

The trial has been extended by 52 weeks. The extension will consist of two 26-week periods:

1. Week 27-52 after randomisation

   - All subjects will continue receiving sitagliptin or liraglutide at unchanged dose and dosing regimen.
2. Week 53-78 after randomisation

   * Subjects receiving sitagliptin at the end of week 52 after randomisation will discontinue sitagliptin and will be randomised 1:1 to liraglutide 1.2 mg/day or liraglutide 1.8 mg/day. Liraglutide will be initiated at a dose of 0.6 mg/day, and increased to 1.2 mg/day or 1.8 mg/day in weekly intervals.
   * Subjects receiving liraglutide 1.2 mg/day or 1.8 mg/day at the end of week 52 after randomisation will continue the treatment at unchanged dose and dosing regimen. Trial completion is planned for June 2010.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treatment with metformin alone for at least three months
* HbA1c (glycosylated haemoglobin A1c) 7.5-10.0% (both inclusive)
* Body Mass Index (BMI) less than or equal to 45.0

Exclusion Criteria:

* Previous treatment with insulin, glucagon like peptide-1 (GLP-1) receptor agonists or dipeptidyl peptidase-4 (DPP-4) inhibitors
* Treatment with anti-diabetic drugs other than metformin within the last three months
* Any serious medical condition
* Females who are pregnant, have the intention of becoming pregnant or are breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (152):
- United States (57):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Crystal River, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Saint Cloud, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Lithia Springs, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Cleveland, Mississippi
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Rosedale, New York
  - Novo Nordisk Investigational Site, Pinehurst, North Carolina
  - Novo Nordisk Investigational Site, Tabor City, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Cuyahoga Falls, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Eugene, Oregon
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, New Braunfels, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (8):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Newmarket, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Hamilton
- Croatia (3):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Sisak
  - Novo Nordisk Investigational Site, Slavonski Brod
- France (8):
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Limoges
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Saint-Mandé
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (12):
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Herrenberg
  - Novo Nordisk Investigational Site, Kassel
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Riesa
  - Novo Nordisk Investigational Site, Schönebeck
  - Novo Nordisk Investigational Site, Ulm
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wangen
- Novo Nordisk Investigational Site, Dublin, Ireland
- Italy (9):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Messina
  - Novo Nordisk Investigational Site, Olbia
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Pavia
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Siena
  - Novo Nordisk Investigational Site, Trieste
- Netherlands (10):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Beek
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Hengelo
  - Novo Nordisk Investigational Site, Leiden
  - Novo Nordisk Investigational Site, Roelofarendsveen
  - Novo Nordisk Investigational Site, Stadskanaal
  - Novo Nordisk Investigational Site, Zevenaar
  - Novo Nordisk Investigational Site, Zoetermeer
- Puerto Rico (5):
  - Novo Nordisk Investigational Site, Caquas
  - Novo Nordisk Investigational Site, Guaynabo
  - Novo Nordisk Investigational Site, Manatí
  - Novo Nordisk Investigational Site, Rio Piedras
  - Novo Nordisk Investigational Site, Trujillo Alto
- Romania (4):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Craiova, Dolj
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Timișoara
- Serbia and Montenegro (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Nis
- Slovakia (3):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Nitra
  - Novo Nordisk Investigational Site, Nové Zámky
- Slovenia (3):
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Novo Mesto
  - Novo Nordisk Investigational Site, Trbovlje
- Spain (8):
  - Novo Nordisk Investigational Site, Alzira
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Getafe
  - Novo Nordisk Investigational Site, L'Hospitalet de Llobregat
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Oviedo
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Puerto del Rosario
- United Kingdom (19):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Abergavenny
  - Novo Nordisk Investigational Site, Aldershot
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Chippenham
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Letchworth Garden City
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Maidstone
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Pratley RE, Nauck M, Bailey T, Montanya E, Cuddihy R, Filetti S, Thomsen AB, Sondergaard RE, Davies M; 1860-LIRA-DPP-4 Study Group. Liraglutide versus sitagliptin for patients with type 2 diabetes who did not have adequate glycaemic control with metformin: a 26-week, randomised, parallel-group, open-label trial. Lancet. 2010 Apr 24;375(9724):1447-56. doi: 10.1016/S0140-6736(10)60307-8. PMID 20417856
- [Result] Davies M, Pratley R, Hammer M, Thomsen AB, Cuddihy R. Liraglutide improves treatment satisfaction in people with Type 2 diabetes compared with sitagliptin, each as an add on to metformin. Diabet Med. 2011 Mar;28(3):333-7. doi: 10.1111/j.1464-5491.2010.03074.x. PMID 21309842
- [Result] Pratley R, Nauck M, Bailey T, Montanya E, Cuddihy R, Filetti S, Garber A, Thomsen AB, Hartvig H, Davies M; 1860-LIRA-DPP-4 Study Group. One year of liraglutide treatment offers sustained and more effective glycaemic control and weight reduction compared with sitagliptin, both in combination with metformin, in patients with type 2 diabetes: a randomised, parallel-group, open-label trial. Int J Clin Pract. 2011 Apr;65(4):397-407. doi: 10.1111/j.1742-1241.2011.02656.x. Epub 2011 Mar 1. PMID 21355967
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Davies MJ, Chubb BD, Smith IC, Valentine WJ. Cost-utility analysis of liraglutide compared with sulphonylurea or sitagliptin, all as add-on to metformin monotherapy in Type 2 diabetes mellitus. Diabet Med. 2012 Mar;29(3):313-20. doi: 10.1111/j.1464-5491.2011.03429.x. PMID 21883438
- [Result] Pratley RE, Nauck MA, Bailey T, Montanya E, Filetti S, Garber AJ, Thomsen AB, Furber S, Davies M; 1860-LIRA-DPP-4 Study Group. Efficacy and safety of switching from the DPP-4 inhibitor sitagliptin to the human GLP-1 analog liraglutide after 52 weeks in metformin-treated patients with type 2 diabetes: a randomized, open-label trial. Diabetes Care. 2012 Oct;35(10):1986-93. doi: 10.2337/dc11-2113. Epub 2012 Jul 30. PMID 22851600
- [Result] Lee WC, Samyshkin Y, Langer J, Palmer JL. Long-term clinical and economic outcomes associated with liraglutide versus sitagliptin therapy when added to metformin in the treatment of type 2 diabetes: a CORE Diabetes Model analysis. J Med Econ. 2012;15 Suppl 2:28-37. doi: 10.3111/13696998.2012.716111. Epub 2012 Aug 13. PMID 22834986
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Result] Davidson JA, Orsted DD, Campos C. Efficacy and safety of liraglutide, a once-daily human glucagon-like peptide-1 analogue, in Latino/Hispanic patients with type 2 diabetes: post hoc analysis of data from four phase III trials. Diabetes Obes Metab. 2016 Jul;18(7):725-8. doi: 10.1111/dom.12653. Epub 2016 Apr 28. PMID 26936426
- [Derived] Langer J, Hunt B, Valentine WJ. Evaluating the short-term cost-effectiveness of liraglutide versus sitagliptin in patients with type 2 diabetes failing metformin monotherapy in the United States. J Manag Care Pharm. 2013 Apr;19(3):237-46. doi: 10.18553/jmcp.2013.19.3.237. PMID 23537458
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 158 centres in 13 countries participated: Canada (11), Croatia (3), Germany (12), Ireland (5), Italy (8), Netherlands (8), Romania (4), Serbia (3), Slovakia (6), Slovenia (3), Spain (9), United Kingdom (20) and United States (66). Of the 158 sites approved by an Independent Ethics Committee, 151 actively screened and enrolled subjects.
Pre-assignment Details: Between screening and randomisation, eligible subjects were to continue their usual pre-study metformin dose and dosing frequency.
Period: Week 0-26 (Main Period)
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Started | 225 (Randomised) | 221 (Randomised) | 219 (Randomised) | 0 | 0
Exposed | 221 (4 subjects withdrew before exposure to trial drug and were not included in Full Analysis Set (FAS)) | 218 (3 subjects withdrew before exposure to trial drug and were not included in Full Analysis Set (FAS)) | 219 | 0 | 0
Completed | 169 | 191 | 194 | 0 | 0
Not Completed | 56 | 30 | 25 | 0 | 0
Not completed — Adverse Event | 14 | 15 | 4 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 4 | 0 | 0
Not completed — Protocol Violation | 14 | 4 | 4 | 0 | 0
Not completed — Withdrawal criteria | 10 | 7 | 5 | 0 | 0
Not completed — Unclassified | 14 | 4 | 8 | 0 | 0
Period: Week 26-52 (Extension Period 1)
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Started | 155 (Subjects withdrew before entry to extension period 1) | 176 (Subjects withdrew before entry to extension period 1) | 166 (Subjects withdrew before entry to extension period 1) | 0 | 0
Completed | 135 | 150 | 151 | 0 | 0
Not Completed | 20 | 26 | 15 | 0 | 0
Not completed — Adverse Event | 5 | 10 | 3 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 7 | 0 | 0
Not completed — Withdrawal criteria | 6 | 8 | 2 | 0 | 0
Not completed — Unclassified | 4 | 3 | 1 | 0 | 0
Period: Week 52-78 (Extension Period 2)
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Started | 134 (Subject withdrew before entry to extension period 2) | 150 | 0 (Re-randomised to lira 1.2 or 1.8 mg) | 67 (Re-randomised from sita treatment group. Some subjects withdrew before entry to extension period 2.) | 68 (Re-randomised from sita treatment group. Some subjects withdrew before entry to extension period 2.)
Completed | 124 | 135 | 0 | 59 | 63
Not Completed | 10 | 15 | 0 | 8 | 5
Not completed — Adverse Event | 0 | 3 | 0 | 6 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 1 | 1
Not completed — Lack of Efficacy | 3 | 3 | 0 | 0 | 0
Not completed — Withdrawal criteria | 4 | 3 | 0 | 1 | 3
Not completed — Unclassified | 2 | 4 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg | Total
Number analyzed (Participants) | 225 | 221 | 219 | 0 | 0 | 665
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.6) | 55.0 (9.1) | 55.0 (9.0) |  |  | 55.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 105 | 99 |  |  | 313
  Male | 116 | 116 | 120 |  |  | 352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 34 | 35 |  |  | 108
  Not Hispanic or Latino | 186 | 187 | 184 |  |  | 557
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 |  |  | 3
  Asian | 6 | 4 | 1 |  |  | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 |  |  | 2
  Black or African American | 22 | 16 | 10 |  |  | 48
  White | 184 | 193 | 199 |  |  | 576
  More than one race | 0 | 0 | 0 |  |  | 0
  Unknown or Not Reported | 9 | 8 | 8 |  |  | 25
Body Mass Index (BMI) at Screening [Mean (Standard Deviation); unit: kg/m^2] | 32.6 (5.2) | 33.1 (5.1) | 32.6 (5.4) |  |  | 32.8 (5.2)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — The time (in years) the patient had been diagnosed with diabetes when screened for the trial
  years | 6.0 (4.5) | 6.4 (5.4) | 6.3 (5.4) |  |  | 6.2 (5.1)
Fasting Plasma Glucose (FPG) at Randomisation [Mean (Standard Deviation); unit: mmol/L] | 10.1 (2.4) | 9.9 (2.4) | 10.0 (2.0) |  |  | 10.0 (2.3)
Glycosylated Haemoglobin A1c (HbA1c) at Randomisation [Mean (Standard Deviation); unit: Percentage point of total HbA1c] | 8.4 (0.8) | 8.4 (0.7) | 8.5 (0.7) |  |  | 8.4 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) at Week 26
Description: Calculated as an estimate of the mean change from baseline in glycosylated haemoglobin A1c (HbA1c) at Week 26.
Time Frame: Week 0, Week 26
Population: FAS (full analysis set) using LOCF (last observation carried forward) is all randomised subjects who had been exposed to at least one dose of trial drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 210 | 0 | 0
Percentage point of total HbA1c | -1.24 (0.07) | -1.5 (0.06) | -0.9 (0.07) |  |
Statistical Analysis 1: Comparison: Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg vs Sita -> Sita; ANCOVA with treatment and country as fixed effects and baseline HbA1c as covariate. Hieracheal testing of non-inferiority followed by superiority; Test type: Non-Inferiority or Equivalence — Non-inferiority concluded if upper confidence interval of test was below 0.4%. Superiority concluded if upper limit of confidence interval was below 0%; p = 0.0001, ANCOVA — Multiple comparisons not applicable due to the hieracheal testing; Adjusted for treatment and country (fixed effects) and baseline HbA1c (covariate); Estimated treatment difference, LS Mean = -0.6, 95% CI [-0.77 to -0.43]
Statistical Analysis 2: Comparison: Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg vs Sita -> Sita; ANCOVA with treatment and country as fixed effects and baseline HbA1c as covariate. Hieracheal testing of non-inferiority followed by superiority. Liraglutide 1.2 mg versus sitagliptin only tested if liraglutide 1.8 mg was superior to sitagliptin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANCOVA — Multiple comparisons not applicable due to the hieracheal testing; Adjusted for treatment and country (fixed effects) and baseline HbA1c (covariate); Estimated treatment difference, LS Mean = -0.34, 95% CI [-0.51 to -0.16]

2. Primary Outcome: Mean Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) at Week 52
Description: Calculated as an estimate of the mean change from baseline in glycosylated haemoglobin A1c (HbA1c) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 210 | 0 | 0
Percentage point of total HbA1c | -1.29 (0.07) | -1.51 (0.07) | -0.88 (0.07) |  |
Statistical Analysis 1: Comparison: Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg vs Sita -> Sita; ANCOVA with treatment and country as fixed effects and baseline HbA1c as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANCOVA — Multiple comparisons not applicable due to the hieracheal testing; Adjusted for treatment and country (fixed effects) and baseline HbA1c (covariate); Estimated Treatment Difference, LS Mean = -0.63, 95% CI [-0.81 to -0.44] — Lira 1.8 - Sita
Statistical Analysis 2: Comparison: Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg vs Sita -> Sita; ANCOVA with treatment and country as fixed effects and baseline HbA1c as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANCOVA — Multiple comparisons not applicable due to the hieracheal testing; Adjusted for treatment and country (fixed effects) and baseline HbA1c (covariate); Estimated Treatment Difference, LS Mean = -0.40, 95% CI [-0.59 to -0.22] — Lira 1.2 - Sita

3. Primary Outcome: Mean Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) at Week 78
Description: Calculated as an estimate of the mean change from baseline in glycosylated haemoglobin A1c (HbA1c) at Week 78.
Time Frame: Week 0, Week 78
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 0 | 0 | 0
Percentage point of total HbA1c | -0.94 (0.08) | -1.28 (0.07) |  |  |

4. Primary Outcome: Mean Change in Glycosylated Haemoglobin A1c (HbA1c) From Week 52 to Week 78
Description: Mean Change in Glycosylated Haemoglobin A1c (HbA1c) from Week 52 to Week 78
Time Frame: Week 52, Week 78
Population: Extension 2 FAS using LOCF (last observation carried forward) is all subjects in the FAS who completed 52 weeks of treatment and who were exposed in the last extension period (week 52 to week 78)
Measure: Mean (Standard Deviation); unit: Percentage point of total HbA1c
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
Percentage point of total HbA1c |  |  |  | -0.24 (0.7) | -0.45 (0.9)
Statistical Analysis 1: Comparison: Sita -> Sita -> Lira 1.2 mg; The t-test was performed to examine whether the change in HbA1c from week 52 to week 78 were different from 0 within each treatment group; Test type: Superiority or Other; p = 0.0060, paired t-test — Multiple comparisons is not applicable; The analysis is not a controlled comparison, and there are no adjustments; Change within treatment group = -0.24, 95% CI [-0.41 to -0.07], Standard Deviation 0.7
Statistical Analysis 2: Comparison: Sita -> Sita -> Lira 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, paired t-test — Multiple comparisons is not applicable; The analysis is not a controlled comparison, and there are no adjustments; Change within treatment group = -0.45, 95% CI [-0.67 to -0.23], Standard Deviation 0.9

5. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c < 7.0% at Week 26
Description: Calculated as the percentage of subjects achieving treatment target of HbA1c < 7.0% at Week 26
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
percentage of subjects | 43 | 55 | 22 |  |

6. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c < 7.0% at Week 52
Description: Calculated as an estimate of the percentage of subjects achieving treatment target of HbA1c < 7.0% at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 210 | 0 | 0
percentage of subjects | 50 | 63 | 27 |  |

7. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c < 7.0% at Week 78
Description: Calculated as an estimate of the percentage of subjects achieving treatment target of HbA1c < 7.0% at Week 78. Based on the FAS.
Time Frame: Week 0, Week 78
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 0 | 0 | 0
percentage of subjects | 35 | 51 |  |  |

8. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c < 7.0% at Week 78
Description: Calculated as an estimate of the percentage of subjects achieving treatment target of HbA1c < 7.0% at Week 78. Based on the extension 2 FAS.
Time Frame: Week 0, Week 78
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
percentage of subjects |  |  |  | 49 | 50

9. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c =< 6.5% at Week 26
Description: Calculated as the percentage of subjects achieving treatment target of HbA1c =< 6.5% at Week 26
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
percentage of subjects | 23 | 36 | 12 |  |

10. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c =< 6.5% at Week 52
Description: Calculated as an estimate of the percentage of subjects achieving treatment target of HbA1c =< 6.5% at Week 52
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 210 | 0 | 0
percentage of subjects | 24 | 40 | 17 |  |

11. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c =< 6.5% at Week 78
Description: Calculated as an estimate of the percentage of subjects achieving treatment target of HbA1c =< 6.5% at Week 78. Based on the FAS.
Time Frame: Week 0, Week 78
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 211 | 214 | 0 | 0 | 0
percentage of subjects | 12 | 27 |  |  |

12. Secondary Outcome: Percentage of Subjects Achieving Treatment Target of HbA1c =< 6.5% at Week 78
Description: Calculated as an estimate of the percentage of subjects achieving treatment target of HbA1c =< 6.5% at Week 78. Based on the extension 2 FAS.
Time Frame: Week 0, Week 78
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
percentage of subjects |  |  |  | 29 | 25

13. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 26
Description: Calculated as an estimate of the mean change from baseline in body weight at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 215 | 214 | 215 | 0 | 0
kg | -2.86 (0.27) | -3.38 (0.27) | -0.96 (0.27) |  |

14. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 52
Description: Calculated as an estimate of the mean change from baseline in body weight at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 215 | 214 | 215 | 0 | 0
kg | -2.78 (0.31) | -3.68 (0.31) | -1.16 (0.31) |  |

15. Secondary Outcome: Mean Change in Body Weight From Week 52 to Week 78
Description: Mean change in body weight from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
kg |  |  |  | -1.64 (3) | -2.48 (3.6)

16. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: Calculated as an estimate of the mean change from baseline in fasting plasma glucose (FPG) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 212 | 210 | 0 | 0
mmol/L | -1.87 (0.15) | -2.14 (0.15) | -0.83 (0.15) |  |

17. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: Calculated as an estimate of the mean change from baseline in fasting plasma glucose (FPG) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 212 | 209 | 0 | 0
mmol/L | -1.71 (0.17) | -2.04 (0.17) | -0.59 (0.17) |  |

18. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 78
Description: Calculated as an estimate of the mean change in fasting plasma glucose (FPG) from baseline to Week 78.
Time Frame: Week 0, Week 78
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 212 | 0 | 0 | 0
mmol/L | -1.30 (0.18) | -1.65 (0.18) |  |  |

19. Secondary Outcome: Mean Change in Fasting Plasma Glucose (FPG) From Week 52 to Week 78
Description: Mean change in fasting plasma glucose (FPG) Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 65 | 67
mmol/L |  |  |  | -0.84 (1.8) | -1.42 (2.1)

20. Secondary Outcome: Mean Change From Baseline in Beta-cell Function at Week 26
Description: Calculated as an estimate of the mean change from baseline in beta-cell function at Week 26.
  Derived from fasting plasma glucose (FPG) and fasting insulin using the homeostatic model assessment (HOMA) method with the assumption that normal-weight subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 196 | 208 | 201 | 0 | 0
percentage point | 27.23 (3.82) | 28.70 (3.75) | 4.18 (3.79) |  |

21. Secondary Outcome: Mean Change From Baseline in Beta-cell Function at Week 52
Description: Calculated as an estimate of the mean change from baseline in beta-cell function at Week 52.
  Derived from fasting plasma glucose (FPG) and fasting insulin using the homeostatic model assessment (HOMA) method with the assumption that normal-weight subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 196 | 208 | 200 | 0 | 0
percentage point | 22.58 (3.31) | 25.76 (3.25) | 3.98 (3.30) |  |

22. Secondary Outcome: Mean Change in Beta-cell Function From Week 52 to Week 78
Description: Mean change in beta-cell function from Week 52 to Week 78. Derived from fasting plasma glucose (FPG) and fasting insulin using the homeostatic model assessment (HOMA) method with the assumption that normal-weight subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage point
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 64 | 64
percentage point |  |  |  | 13.31 (29.4) | 23.09 (43.7)

23. Secondary Outcome: Mean Change From Baseline in Total Cholesterol at Week 26
Description: Calculated as an estimate of the mean change from baseline in total cholesterol at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 194 | 202 | 201 | 0 | 0
mmol/L | -0.03 (0.06) | -0.17 (0.05) | -0.02 (0.05) |  |

24. Secondary Outcome: Mean Change From Baseline in Total Cholesterol at Week 52
Description: Calculated as an estimate of the mean change from baseline in total cholesterol at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 195 | 203 | 200 | 0 | 0
mmol/L | -0.01 (0.06) | -0.09 (0.06) | 0.03 (0.06) |  |

25. Secondary Outcome: Mean Change in Total Cholesterol From Week 52 to Week 78
Description: Mean change in total cholesterol from Week 52 to Week 78
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 65 | 67
mmol/L |  |  |  | -0.16 (0.8) | -0.24 (0.7)

26. Secondary Outcome: Mean Change From Baseline in Low-density Lipoprotein-cholesterol (LDL-C) at Week 26
Description: Calculated as an estimate of the mean change in low-density lipoprotein-cholesterol (LDL-C) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 194 | 202 | 200 | 0 | 0
mmol/L | 0.08 (0.05) | 0.05 (0.05) | 0.13 (0.05) |  |

27. Secondary Outcome: Mean Change From Baseline in Low-density Lipoprotein-cholesterol (LDL-C) at Week 52
Description: Calculated as an estimate of the mean change in low-density lipoprotein-cholesterol (LDL-C) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 195 | 203 | 199 | 0 | 0
mmol/L | 0.09 (0.05) | 0.09 (0.05) | 0.17 (0.05) |  |

28. Secondary Outcome: Mean Change in Low-density Lipoprotein-cholesterol (LDL-C) From Week 52 to Week 78
Description: Mean change in low-density lipoprotein-cholesterol (LDL-C) from week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 65 | 67
mmol/L |  |  |  | -0.22 (0.7) | -0.25 (0.6)

29. Secondary Outcome: Mean Change From Baseline in High-density Lipoprotein-cholesterol (HDL-C) at Week 26
Description: Calculated as an estimate of the mean change from baseline in high-density lipoprotein-cholesterol (HDL-C) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 194 | 201 | 201 | 0 | 0
mmol/L | 0.00 (0.01) | 0.00 (0.01) | 0.00 (0.01) |  |

30. Secondary Outcome: Mean Change From Baseline in High-density Lipoprotein-cholesterol (HDL-C) at Week 52
Description: Calculated as an estimate of the mean change from baseline in high-density lipoprotein-cholesterol (HDL-C) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 195 | 202 | 200 | 0 | 0
mmol/L | 0.01 (0.01) | 0.02 (0.01) | 0.01 (0.01) |  |

31. Secondary Outcome: Mean Change in High-density Lipoprotein-cholesterol (HDL-C) From Week 52 to Week 78
Description: Mean change in high-density lipoprotein-cholesterol (HDL-C) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 65 | 67
mmol/L |  |  |  | 0.02 (0.1) | -0.01 (0.2)

32. Secondary Outcome: Mean Change From Baseline in Very Low-density Lipoprotein-cholesterol (VLDL-C) at Week 26
Description: Calculated as an estimate of the change from baseline in very low-density lipoprotein-cholesterol (VLDL-C) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 194 | 201 | 199 | 0 | 0
mmol/L | -0.11 (0.03) | -0.20 (0.03) | -0.15 (0.03) |  |

33. Secondary Outcome: Mean Change From Baseline in Very Low-density Lipoprotein-cholesterol (VLDL-C) at Week 52
Description: Calculated as an estimate of the change from baseline in very low-density lipoprotein-cholesterol (VLDL-C) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 195 | 202 | 198 | 0 | 0
mmol/L | -0.11 (0.04) | -0.19 (0.04) | -0.15 (0.04) |  |

34. Secondary Outcome: Mean Change in Very Low-density Lipoprotein-cholesterol (VLDL-C) at Week 52 to Week 78
Description: Mean change in very low-density lipoprotein-cholesterol (VLDL-C) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 65 | 67
mmol/L |  |  |  | 0.03 (0.3) | 0.02 (0.3)

35. Secondary Outcome: Mean Change From Baseline in Triglycerides (TG) at Week 26
Description: Calculated as an estimate of the change from baseline in triglycerides (TG) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 191 | 199 | 198 | 0 | 0
mmol/L | -0.19 (0.10) | -0.43 (0.09) | -0.40 (0.09) |  |

36. Secondary Outcome: Mean Change From Baseline in Triglycerides (TG) at Week 52
Description: Calculated as an estimate of the change from baseline in triglycerides (TG) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 194 | 200 | 197 | 0 | 0
mmol/L | -0.10 (0.10) | -0.32 (0.10) | -0.23 (0.10) |  |

37. Secondary Outcome: Mean Change in Triglycerides (TG) From Week 52 to Week 78
Description: Mean change in triglycerides (TG) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 64 | 66
mmol/L |  |  |  | -0.20 (0.8) | -0.26 (0.8)

38. Secondary Outcome: Mean Change From Baseline in Free Fatty Acids (FFA) at Week 26
Description: Calculated as an estimate of the change from baseline in free fatty acids (FFA) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 147 | 149 | 158 | 0 | 0
mmol/L | -0.03 (0.02) | -0.07 (0.02) | -0.05 (0.02) |  |

39. Secondary Outcome: Mean Change From Baseline in Free Fatty Acids (FFA) at Week 52
Description: Calculated as an estimate of the change from baseline in free fatty acids (FFA) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 170 | 177 | 176 | 0 | 0
mmol/L | -0.07 (0.02) | -0.10 (0.02) | -0.06 (0.02) |  |

40. Secondary Outcome: Mean Change in Free Fatty Acids (FFA) From Week 52 to Week 78
Description: Mean change in free fatty acids (FFA) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 60 | 65
mmol/L |  |  |  | 0.02 (0.3) | -0.01 (0.3)

41. Secondary Outcome: Mean Change From Baseline in Apolipoprotein B at Week 26
Description: Calculated as an estimate of the change from baseline in apolipoprotein B (ApoB) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 164 | 175 | 182 | 0 | 0
g/L | -0.06 (0.01) | -0.07 (0.01) | -0.05 (0.01) |  |

42. Secondary Outcome: Mean Change From Baseline in Apolipoprotein B at Week 52
Description: Calculated as an estimate of the change from baseline in apolipoprotein B (ApoB) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 184 | 192 | 195 | 0 | 0
g/L | -0.03 (0.01) | -0.03 (0.01) | -0.03 (0.01) |  |

43. Secondary Outcome: Mean Change in Apolipoprotein B From Week 52 to Week 78
Description: Mean change in apolipoprotein B (ApoB) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 66 | 68
mmol/L |  |  |  | 0.23 (0.4) | 0.17 (0.4)

44. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C-reactive Protein (hsCRP) at Week 26
Description: Calculated as an estimate of the mean change from baseline in highly sensitive C-reactive protein (hsCRP) at week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 205 | 209 | 205 | 0 | 0
mg/L | -1.02 (0.31) | -0.99 (0.31) | -0.66 (0.31) |  |

45. Secondary Outcome: Mean Change From Baseline in Plasminogen Activator Inhibitor-1 (PAI-1) at Week 26.
Description: Calculated as an estimate of the mean change from baseline in plasminogen activator inhibitor-1 (PAI-1) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 188 | 198 | 182 | 0 | 0
U/L | -833 (945.1) | -561 (941.1) | 586 (952) |  |

46. Secondary Outcome: Mean Change From Baseline in Interleukin-6 (IL-6) at Week 26.
Description: Calculated as an estimate of the mean change from baseline in interleukin-6 (IL-6) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 204 | 210 | 206 | 0 | 0
pg/mL | -1.70 (2.49) | 1.71 (2.47) | 0.91 (2.49) |  |

47. Secondary Outcome: Mean Change From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) at Week 26.
Description: Calculated as an estimate of the mean change from baseline in N-terminal pro B-type Natriuretic Peptide (NT-proBNP) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 204 | 209 | 205 | 0 | 0
pmol/L | 5.19 (2.07) | 3.74 (2.06) | 3.71 (2.07) |  |

48. Secondary Outcome: Mean Change From Baseline in Adiponectin at Week 26.
Description: Calculated as an estimate of the mean change from baseline in Adiponectin at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcg/mL
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 202 | 210 | 207 | 0 | 0
mcg/mL | 1.69 (0.19) | 1.51 (0.19) | 1.35 (0.19) |  |

49. Secondary Outcome: Mean Change From Baseline in Tumour Necrosis Factor Alpha (TNF-alpha) at Week 26.
Description: Calculated as an estimate of the mean change from baseline in Tumour Necrosis Factor Alpha (TNF-alpha) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 195 | 204 | 196 | 0 | 0
pg/mL | -0.55 (0.25) | -0.74 (0.25) | -0.53 (0.25) |  |

50. Secondary Outcome: Mean Change From Baseline in Von Willebrand Factor (vWf) at Week 26.
Description: Calculated as an estimate of the mean change from baseline in von Willebrand Factor (vWf) at Week 26. vWf is a blood glycoprotein involved in haemostasis.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 189 | 193 | 183 | 0 | 0
percentage point | -1.73 (2.77) | -4.34 (2.76) | -1.8 (2.82) |  |

51. Secondary Outcome: Mean Change From Baseline in Waist to Hip Ratio at Week 26.
Description: Calculated as an estimate of the mean change from baseline in Waist to Hip Ratio at Week 26. The measure is assessed as the circumference of the waist divided by the circumference of the hip.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/cm
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 208 | 207 | 0 | 0
cm/cm | -0.01 (0.00) | -0.01 (0.00) | -0.00 (0.00) |  |

52. Secondary Outcome: Mean Change From Baseline in Waist to Hip Ratio at Week 52
Description: Calculated as an estimate of the mean change from baseline in Waist to Hip Ratio at Week 52. The measure is assessed as the circumference of the waist divided by the circumference of the hip.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/cm
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 208 | 207 | 0 | 0
cm/cm | -0.00 (0.00) | -0.01 (0.00) | -0.00 (0.00) |  |

53. Secondary Outcome: Mean Change in Waist to Hip Ratio From Week 52 to Week 78
Description: Mean change in Waist to Hip Ratio from Week 52 to Week 78. The measure is assessed as the circumference of the waist divided by the circumference of the hip.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm/cm
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 66 | 67
cm/cm |  |  |  | -0.01 (0) | -0.00 (0)

54. Secondary Outcome: Mean Change From Baseline in Waist Circumference at Week 26.
Description: Calculated as an estimate of the mean change from baseline in Waist Circumference at Week 26
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 208 | 208 | 0 | 0
cm | -2.69 (0.35) | -2.63 (0.36) | -1.12 (0.36) |  |

55. Secondary Outcome: Mean Change From Baseline in Waist Circumference at Week 52
Description: Calculated as an estimate of the mean change from baseline in Waist Circumference at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: participants
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 210 | 208 | 208 | 0 | 0
participants | -2.36 (0.38) | -3.02 (0.38) | -1.23 (0.38) |  |

56. Secondary Outcome: Mean Change in Waist Circumference From Week 52 to Week 78
Description: Mean change in Waist Circumference from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 66 | 68
kg |  |  |  | -1.33 (3.5) | -2.05 (4.1)

57. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) at Week 26
Description: Calculated as an estimate of the mean change from baseline in Systolic Blood Pressure (SBP) at Week 26
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 213 | 214 | 213 | 0 | 0
mmHg | -0.55 (0.89) | -0.72 (0.89) | -0.94 (0.89) |  |

58. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) at Week 52
Description: Calculated as an estimate of the mean change from baseline in systolic blood pressure (SBP) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 213 | 214 | 213 | 0 | 0
mmHg | -0.37 (0.93) | -2.55 (0.93) | -1.03 (0.93) |  |

59. Secondary Outcome: Mean Change in Systolic Blood Pressure (SBP) From Week 52 to Week 78
Description: Mean change in systolic blood pressure (SBP) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
mmHg |  |  |  | -2.12 (14.6) | 0.35 (12.4)

60. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (DBP) at Week 26
Description: Calculated as an estimate of the mean change from baseline in diastolic blood pressure (DBP) at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 213 | 214 | 213 | 0 | 0
mmHg | -0.71 (0.60) | 0.07 (0.59) | -1.78 (0.60) |  |

61. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (DBP) at Week 52
Description: Calculated as an estimate of the mean change from baseline in diastolic blood pressure (DBP) at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 213 | 214 | 213 | 0 | 0
mmHg | -0.53 (0.57) | -0.87 (0.57) | -1.47 (0.57) |  |

62. Secondary Outcome: Mean Change in Diastolic Blood Pressure (DBP) From Week 52 to Week 78
Description: Mean change in diastolic blood pressure (DBP) from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
mmHg |  |  |  | -0.60 (10.0) | 0.03 (8.9)

63. Secondary Outcome: Mean Change From Baseline in Pulse at Week 26
Description: Calculated as an estimate of the mean change from baseline in pulse at Week 26.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats/minute
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 212 | 214 | 211 | 0 | 0
beats/minute | 2.32 (0.59) | 3.94 (0.58) | -0.64 (0.59) |  |

64. Secondary Outcome: Mean Change From Baseline in Pulse at Week 52
Description: Calculated as an estimate of the mean change from baseline in pulse at Week 52.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 212 | 214 | 211 | 0 | 0
mmHg | 1.72 (0.60) | 3.09 (0.60) | 0.09 (0.60) |  |

65. Secondary Outcome: Mean Change in Pulse From Week 52 to Week 78
Description: Mean change in pulse from Week 52 to Week 78.
Time Frame: Week 52, Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 67 | 68
beats/minute |  |  |  | 0.90 (8.4) | 2.19 (7.7)

66. Secondary Outcome: Mean Change From Baseline in Overall Treatment Satisfaction (OTS) at Week 26
Description: The Overall Treatment Satisfaction is a sum of 6 items from the Diabetes Treatment Satisfaction Questionnaire, which is a self-assessment of treatment satisfaction. The scale of each sub-item goes from 0 (lowest satisfaction) to 6 (highest satisfaction) and the overall scale of OTS therefore goes from 0 to 36.
Time Frame: Week 0, Week 26
Population: Patient Reported Outcome Analysis Set consisted of all subjects in the FAS, except subjects from countries Serbia, Slovakia and Slovenia
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 164 | 171 | 170 | 0 | 0
scores on a scale | 3.51 (0.49) | 4.35 (0.48) | 2.96 (0.48) |  |

67. Secondary Outcome: Mean Change From Baseline in Overall Treatment Satisfaction (OTS) at Week 52
Description: as for outcome 66
Time Frame: Week 0, Week 52
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 163 | 165 | 169 | 0 | 0
scores on a scale | 3.32 (0.49) | 4.31 (0.48) | 2.96 (0.48) |  |

68. Secondary Outcome: Mean Change in Overall Treatment Satisfaction (OTS) From Week 52 to Week 78
Description: as for outcome 66
Time Frame: Week 52, Week 78
Population: Extension 2 Patient Reported Outcome Analysis Set consisted of all subjects in the Extension 2 FAS, except subjects from countries Serbia, Slovakia and Slovenia
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 0 | 0 | 0 | 54 | 48
scores on a scale |  |  |  | 1.48 (4.4) | 0.98 (6.1)

69. Secondary Outcome: Hypoglyceamic Episodes, Weeks 0-26
Description: Number of hypoglycaemic episodes from Week 0 to Week 26, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-26
Population: The safety analysis set is all randomised subjects who had been exposed to at least one dose of the trial products.
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
episodes
  Major | 1 | 0 | 0 |  |
  Minor | 17 | 37 | 11 |  |
  Symptoms only | 12 | 15 | 10 |  |
  Unclassified | 0 | 1 | 0 |  |

70. Secondary Outcome: Hypoglycaemic Episodes (Excluding Outlier Subject), Weeks 0-26
Description: as for outcome 69
Time Frame: Weeks 0-26
Population: The safety analysis set is all randomised subjects who had been exposed to at least one dose of the trial products. An outlier subject from the lira 1.8 mg+met group, who experienced 21 minor hypoglycaemic episodes was excluded from this analysis.
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 217 | 219 | 0 | 0
episodes
  Major | 1 | 0 | 0 |  |
  Minor | 17 | 16 | 11 |  |
  Symptoms only | 12 | 15 | 10 |  |
  Unclassified | 0 | 1 | 0 |  |

71. Secondary Outcome: Hypoglyceamic Episodes, Weeks 0-52
Description: Number of hypoglycaemic episodes from Week 0 to Week 52, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-52
Population: The safety analysis set is all randomised subjects who had been exposed to at least one dose of the trial products.
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
episodes
  Major | 1 | 0 | 0 |  |
  Minor | 24 | 51 | 25 |  |
  Symptoms only | 14 | 29 | 12 |  |
  Unclassified | 0 | 1 | 0 |  |

72. Secondary Outcome: Hypoglycaemic Episodes (Excluding Outlier Subject), Weeks 0-52
Description: as for outcome 71
Time Frame: Weeks 0-52
Population: The safety analysis set is all randomised subjects who had been exposed to at least one dose of the trial products. An outlier subject from the lira 1.8 mg+met group, who experienced 23 minor hypoglycaemic episodes was excluded from this analysis.
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
episodes
  Major | 1 | 0 | 0 |  |
  Minor | 24 | 28 | 25 |  |
  Symptoms only | 14 | 29 | 12 |  |
  Unclassified | 0 | 1 | 0 |  |

73. Secondary Outcome: Hypoglyceamic Episodes, Weeks 0-78
Description: Number of hypoglycaemic episodes from Week 0 to Week 78, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-78
Population: The safety analysis set is all randomised subjects who had been exposed to at least one dose of the trial products.
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
episodes
  Major | 2 | 0 | 0 |  |
  Minor | 36 | 56 | 34 |  |
  Symptoms only | 18 | 40 | 13 |  |
  Unclassified | 0 | 1 | 0 |  |

74. Secondary Outcome: Hypoglycaemic Episodes (Excluding Outlier Subject), Weeks 0-78
Description: as for outcome 73
Time Frame: Weeks 0-78
Population: as for outcome 72
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 221 | 218 | 219 | 0 | 0
episodes
  Major | 2 | 0 | 0 |  |
  Minor | 36 | 33 | 34 |  |
  Symptoms only | 18 | 40 | 13 |  |
  Unclassified | 0 | 1 | 0 |  |

75. Secondary Outcome: Hypoglycaamic Episodes, Weeks 52-78
Description: Number of hypoglycaemic episodes from Week 52 to Week 78, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Week 52-78
Population: as for outcome 4
Measure: Number; unit: episodes
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita | Sita -> Sita -> Lira 1.2 mg | Sita -> Sita -> Lira 1.8 mg
Number analyzed (Participants) | 134 | 150 | 0 | 67 | 68
episodes
  Major | 1 | 0 |  | 0 | 0
  Minor | 12 | 5 |  | 3 | 6
  Symptoms only | 3 | 11 |  | 1 | 0
  Unclassified | 0 | 0 |  | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 78 weeks.
Description: The safety analysis set is all randomised subjects who had been exposed to at least one dose of the trial products.
Arm/Group | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg | Sita -> Sita
Serious Adverse Events (participants affected / at risk) | 12/221 | 19/218 | 17/219
Other Adverse Events (participants affected / at risk) | 120/221 | 134/218 | 106/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg (N=221) | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg (N=218) | Sita -> Sita (N=219)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mycetoma mycotic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected sebaceous cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Abcess Limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecytitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoe syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.2 mg -> Lira 1.2 mg -> Lira 1.2 mg (N=221) | Lira 1.8 mg -> Lira 1.8 mg -> Lira 1.8 mg (N=218) | Sita -> Sita (N=219)
Nausea (Gastrointestinal disorders) | 48 (60) | 61 (73) | 36 (45)
Diarrhoea (Gastrointestinal disorders) | 21 (30) | 29 (52) | 24 (40)
Vomiting (Gastrointestinal disorders) | 18 (27) | 24 (28) | 15 (21)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 17 (23) | 11 (17)
Constipation (Gastrointestinal disorders) | 10 (11) | 14 (16) | 10 (11)
Nasopharyngitis (Infections and infestations) | 33 (42) | 36 (52) | 32 (50)
Influenza (Infections and infestations) | 14 (17) | 7 (7) | 9 (13)
Headache (Nervous system disorders) | 23 (36) | 31 (56) | 33 (50)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 12 (12) | 9 (9)
Fatigue (General disorders) | 9 (9) | 13 (14) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 16 (27) | 11 (16) | 14 (20)
Blood calcitonin increased (Investigations) | 9 (9) | 11 (14) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (21) | 14 (16) | 13 (16)
Dizziness (Nervous system disorders) | 10 (10) | 14 (19) | 8 (8)
Hypertension (Vascular disorders) | 13 (13) | 14 (14) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.